CLINICAL TRIAL: NCT04616404
Title: The Metabolic Effects of Cynara Supplementation in Overweight and Obese Class I Subjects With Newly Detected Impaired Fasting Glycaemia: a Double-blind, Placebo-controlled, Randomized Clinical Trial
Brief Title: The Metabolic Effects of Cynara Supplementation in Overweight and Obese Class I Subjects With Newly Detected Impaired Fasting Glycaemia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Collaborators: Indena S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9321/14122018
Record Dates: First submitted 2020-10-13; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Insulin Sensitivity; Obesity; Overweight
Keywords: impaired fasting glucose; Cynara cardunculus; Insulin Sensitivity; Obesity; Overweight
MeSH Terms: conditions — Insulin Resistance; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator)
  Interventions: Dietary Supplement: 500 mg of artichoke extract
- Control Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 500 mg of artichoke extract — Tablets containing 500 mg of artichoke extract (triple standardized to contain caffeoylquinic acids ≥ 5.0%; flavonoids ≥ 1.5%; cynaropicrin ≥ 1.0%, by HPLC)
  Arms: Intervention Group
Other: Placebo — Tablets with no active ingredient
  Arms: Control Group

SUMMARY:
Impaired fasting glucose (IFG) is a condition that precedes diabetes and increases the risk of developing it. Studies support the hypoglycemic effect of Cynara cardunculus (Cs) extracts due to the content of chlorogenic acid, which is a potent inhibitor of glucose 6-phosphate translocase and of dicaffeoylquinic acid derivatives that modulate the activity of alpha-glucosidase. Given this background, we investigated whether a new highly standardized Cs extract could improve glycaemic control, insulin sensitivity and other metabolic parameters (total, HDL and LDL cholesterol, Triglycerides, ApoB, ApoA, waist circumference, Visceral adipose tissue by DXA) in overweight subjects with newly diagnosed IFG.

ELIGIBILITY:
Inclusion Criteria:

* without history of cardiovascular disease (CVD),
* not taking any medication likely to affect glucose or lipid metabolism (oral hypoglycemic agents and statins)
* free of overt liver, renal and thyroid disease

Exclusion Criteria:

* smoking
* drinking more than two standard alcoholic beverages/day (20 g of alcohol/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Changes on glycemia | Day 0, after 1 month and after 2 months

SECONDARY OUTCOMES:
Changes on total cholesterol (mg/dl), HDL (mg/dl), total cholesterol/HLD, LDL (mg/dl), LDL/HDL, triglycerides (mg/dl), ApoA (mg/dl), ApoB (mg/dl), ApoB/ApoA, creatinine (mg/dl) | Day 0, after 1 month and after 2 months
Changes on AST (UI/l), ALT (UI/l), GGT (U/l) | Day 0, after 1 month and after 2 months
Changes on insulin (mcU/ml) and HOMA index | Day 0, after 1 month and after 2 months
Changes on glycated hemoglobin (%) | Day 0, after 1 month and after 2 months
Changes on A1c-Derived Average Glucose (mmol/l) | Day 0, after 1 month and after 2 months
Changes on maximum blood pressure (mmHg), minimum blood pressure (mmHg) | Day 0, after 1 month
Changes on waist circumference (cm) | Day 0, after 1 month
Changes on VAT (g), lean and fat mass (g) | Day 0, after 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda di Servizi alla Persona ''Istituto Santa Margherita'', Pavia, PV, Italy